CLINICAL TRIAL: NCT05777629
Title: Determination of Compliance to Mediterranean Diet, Impacts on Walking and Quality of Life in Multiple Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Nezihe Otay Lule, Principal Investigator, University of Gaziantep
Other Study IDs: nol
Record Dates: First submitted 2023-01-26; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Mediterranean Diet; Quality of Life; Walking
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multiple Sclerosis (MS) is an autoimmune disease characterized by inflammation, demyelination and axon damage. Affecting approximately 2.5 million individuals around the world and seen mostly in young adults, MS can cause different levels of disability in functional activities, cause limitations in social and professional life, and impair quality of life. Multiple sclerosis is thought to be an autoimmune disease that develops on the basis of genetic predisposition and environmental factors. Nutritional habits and physical activity are important environmental factors. These can be effective in the course of MS and change the quality of life. Compatibility of nutrition with the Mediterranean diet and providing adequate physical activity may be beneficial in increasing physical and mental well-being in general, and therefore the quality of life of the person.

In our country, there is not enough information about the ongoing nutritional habits and physical activity levels of MS patients in their daily lives, and quality of life studies are limited. Our limited knowledge on these issues narrows the possibility of movement in an area that can be corrected in MS patients and thus have a positive impact on their quality of life. The aim of this study is to determine compliance with the Mediterranean diet, the tendency to use various nutritional supplements, physical activity habits, walking-related problems and quality of life in MS patients and to evaluate whether there is a significant relationship between these parameters.

DETAILED DESCRIPTION:
Clinical studies examining the effects of various dietary patterns on MS are ongoing, and evidence is still lacking regarding the use of any specific dietary therapy for individuals with MS. In general, individuals living in high-income western countries where the disease is more common; They lead a sedentary life, are less exposed to sunlight, and are fed a high-energy diet rich in animal-derived saturated fats and refined sugar.

The Mediterranean diet is a nutritional model that is universally thought to improve health, and it is known that the Mediterranean diet has beneficial effects in the prevention and treatment of chronic diseases.The major difference between the Mediterranean diet and the Western-style diet is the source and amount of dietary fat and carbohydrates. The Mediterranean diet is rich in foods containing monounsaturated fat (especially omega-3), antioxidant vitamins and minerals (vitamins A, C, E, folic acid, selenium, zinc, calcium), which are thought to have positive effects on the prevention and course of MS.

Preferring vegetable oils instead of animal fats in Mediterranean type diet, preferring fish instead of red meat consumption, preferring low-fat / fat-free milk and dairy products, limiting the intake of simple sugar and refined carbohydrates, increasing the consumption of fruits and vegetables rich in pulp and antioxidants. It is thought that this type of nutrition may positively affect the course and treatment of immune diseases by reducing inflammation.

Although there is no effective clinical evidence for the application of nutritional support as complementary therapy in MS patients, it is known that patients often use various nutritional supplements to reduce symptoms that negatively affect their quality of life. It is also important to determine the frequency of current nutritional support use in order to prevent unconscious use of nutritional support in the group.

Because the most common symptoms of MS are muscle weakness, individuals with MS are often less physically active than age-matched adults

All these negativities result in decreased functional activities, loss of mobility and balance problems.

Walking and, in a broader sense, mobility are functions that are frequently affected in MS and have a high negative impact on quality of life. Gait problems are not uncommon in MS, and it is reported that a significant portion of individuals in this group are adversely affected by their daily living activities.

The aim of this study is to determine compliance with the Mediterranean diet, the tendency to use various nutritional supplements, physical activity habits, walking-related problems and quality of life in MS patients and to evaluate whether there is a significant relationship between these parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Being between the ages of 18-65
2. Having been diagnosed with multiple sclerosis
3. Having voluntarily agreed to participate in the research
4. Absence of exclusion criteria

Exclusion Criteria:

1. Being under the age of 18 and over the age of 65
2. Being pregnant or in the postpartum period during the research
3. Having an attack during the research
4. Active infection
5. Having another disease that prevents him from doing physical activity
6. Having a disease that requires a special diet

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with MS between the ages of 18-65
Sampling Method: Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2021-02-28 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Mediterranean Diet Compliance Status | 1 year
  The 14-item Mediterranean Diet Adaptation Scale (PREDIMED) will be used to determine the adaptation status of individuals to the Mediterranean diet. In this scale, there are a total of 14 questions, 12 of which are about food consumption frequency and 2 are about food consumption habits. The score given for each question is 0 or 1 point. Then the scores are summed and the score is evaluated as ≤5 (low agreement), 6-9 (moderate agreement), and ≥10 (high agreement).
Quality of Life Of Multiple Sclerosis Patients | 1 months
  The quality of life of individuals will be determined by the Multiple Sclerosis International Quality of Life Scale. It is evaluated between 0-124 points in total. An increase in the total score is associated with a higher quality of life.
Impacts on Walking | 2 months
  The 12-item Ms Gait Scale will be used to determine the gait impact. 12-item MS Gait Scale: It is a 12-item questionnaire that questions the effect of walking in MS. The difficulties experienced by individuals during walking activity in the last 2 weeks are questioned. Each item contains 5 points (1; not at all impressed, 5; totally impressed). Lower scores indicate better gait impairment
Expanded Disability Status Scale | 1 year
  The disability status of the patients will be determined using the Expanded Disability Status Scale (EDSS). The EDSS scale measures disability and neurological symptoms in MS patients. A score between 0 and 10 is given on the scale. 0 indicates no disability or disorder, 10 indicates MS-related death

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin EKMEKYAPAR FIRAT, Principal Investigator — Sanko University; Münife NEYAL, Principal Investigator — Sanko University; İpek KATİRCİ KİRMACİ, Principal Investigator — Kahramanmaras Sutcu Imam University; Nezihe OTAY LULE, Principal Investigator — Gaziiantep University
Locations (1):
- UGaziantep, Gaziantep, Turkey (Türkiye)